CLINICAL TRIAL: NCT02334904
Title: Comparison of Aripiprazole Versus Risperidone on Brain Morphology Using MRI
Acronym: CARB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: H14-01075
Record Dates: First submitted 2014-12-12; First posted 2015-01-08 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: First-Episode Psychosis; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be offered the option of taking part in an optional biobanking component of the main study. Eight milliliters of whole blood samples will be collected and stored at -80 degrees Celsius for genotyping to determine if certain genetic polymorphisms predispose individuals to brain changes while taking antipsychotic medications.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aripiprazole: Participants receiving treatment of only aripiprazole, as prescribed to them by their psychiatrists, for a minimum of at least 3 continuous months.
  Interventions: Drug: Aripiprazole
- Risperidone: Participants receiving treatment of only risperidone, as prescribed to them by their psychiatrists, for a minimum of at least 3 continuous months.
  Interventions: Drug: Risperidone
- Controls: Healthy participants who are not taking any antipsychotic medications.

INTERVENTIONS:
Drug: Aripiprazole — To be prescribed and monitored by participant's attending physician (not given to participants as a part of the study)
  Other Names: Abilify
  Groups: Aripiprazole
Drug: Risperidone — To be prescribed and monitored by participant's attending physician (not given to participants as a part of the study).
  Groups: Risperidone

SUMMARY:
Significant changes in brain morphology are observed in people with first-episode psychosis. Studies have shown that total brain volume and particular brain structures are decreased in people with psychosis disorders. Recent evidence suggests that some atypical antipsychotic drugs can maintain or increase brain volumes. Thus, we plan to use MRI scans to measure changes in brain morphology in subjects recently diagnosed with bipolar or psychosis disorders who are taking the atypical antipsychotic drugs aripiprazole or risperidone. Secondary objectives include taking blood samples for fasting metabolic indices and neuropsychiatric measures for comparisons between drug treatments.

DETAILED DESCRIPTION:
The purpose of this study is to use a direct measure of brain volume and matter (by means of MRI) to determine if there is a differential effect between aripiprazole and risperidone on brain morphology in participants with first-episode psychosis. A secondary objective is to see if fasting metabolic indices measured in the blood (i.e. glucose, insulin, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, adiponectin and leptin) are also correlated to changes in brain morphology or symptom severity (as measured by neuropsychiatric assessments).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 12+ years for healthy participants or participants with bipolar disorder; or aged 15+ years for participants with non-affective psychosis.
* Recent admission to the Vancouver/Richmond Early Psychosis Intervention (EPI) program related to first episode psychosis or first episode bipolar disorder;
* Participants being treated with an antipsychotic medication principally for psychosis or for bipolar disorder.
* Participants taking aripiprazole must be taking a dose of at least 10mg/day for the duration of the study.
* Participants must have received a minimum of 3 months of continuous antipsychotic drug treatment with either aripiprazole or risperidone principally for psychosis or bipolar disorder;
* Participants may be in- or outpatients.
* Participants able to give informed consent, or informed consent through legally authorized representative.

Exclusion Criteria:

* Total life time exposure to the antipsychotic drug aripiprazole vs risperidone for less than 3 months at time of consent.
* Previously diagnosed with diabetes mellitus, seizure disorders, mental retardation (IQ < 70), or pregnancy (current or within 3 months postpartum)
* Participants who have been treated/are currently being treated with mood stabilizers (paroxetine, lithium, or valproic acid). Prior or concurrent use of Selective Serotonin Reuptake Inhibitor antidepressants (other than paroxetine) is acceptable..
* Received antipsychotic polypharmacy (treatment with more than one antipsychotic drug)
* Participants who are not able to fluently communicate in English.
* Contraindicated for MRI scan (i.e., has had major surgery in the last 6 months, morbid obesity, claustrophobia, and/or has metal in their bodies from a surgical intervention or working in metalwork, or is unsure if metal is present in their bodies, etc.)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Vancouver.Richmond EPI program who have been on at least 3 months of continuous antipsychotic drug treatment with either aripiprazole or risperidone for first-episode psychosis or bipolar disorder, and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
MRI Brain Scans (Composite Measure) | Day 1 (Visit 1)
  Using structural MRI, we will measure total brain volume (TBV), grey matter volume (GMV), white matter volumes (WMV), and/or volumes of other brain structures.

SECONDARY OUTCOMES:
Metabolic Fasting Blood Work (Composite Measures) | Day 1 (Visit 1)
  By obtaining two tubes of fasting blood, we will determine fasting metabolic parameters of common blood components (lipids, cholesterol, leptin, adiponectin, glucose, and insulin).
Genetic Measures (Composite Measure) | Day 1 (Visit 1)
  An optional component, as obtained from blood work, will be to determine potential genetic variants in several candidate genes (such as BDNF) that predispose some subjects to changes in brain morphology.
Neuropsychological Assessments | At time of Day 1 (Only for those taking antipsychotic medications)
  To assess cognitive functioning for those subject's taking risperidone or aripiprazole, we will administer a set of standard scales and surveys to measure executive and cognitive functioning.
Psychiatric Assessment | At time of Day 1 (Only for those taking antipsychotic medications)
  To assess mental health symptoms for those subject's taking risperidone or aripiprazole, we will administer a set of interviews (PANSS and MINI) to assess mental health symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair M Barr, Ph.D, Principal Investigator — University of British Columbia; Lili Kopala, M.D., Principal Investigator — University of British Columbia
Locations (1):
- BC Mental Health & Addictions Research Institute, Vancouver, British Columbia, Canada